CLINICAL TRIAL: NCT04727801
Title: A Clinical Data Collection Study of Verily Patch
Status: Terminated | Type: Observational
Why Stopped: Decision by the Sponsor
Sponsor: Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 102782
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Febrile; Afebrile
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Febrile (n=50): Febrile is defined as having sublingual temperatures of 37.5 °C or above. All subjects will wear the Verily Patch in the axillary region for up to 8 days. In addition, subjects will measure oral and axillary temperatures using a commercially available thermometer.
  Interventions: Device: Verily Patch
- Afebrile (n=50): Afebrile is defined as having sublingual temperatures of less than 37.5 °C. All subjects will wear the Verily Patch in the axillary region for up to 8 days. In addition, subjects will measure oral and axillary temperatures using a commercially available thermometer.
  Interventions: Device: Verily Patch

INTERVENTIONS:
Device: Verily Patch — The Verily Patch is an investigational wearable temperature sensor that consists of a Patch (Verily Patch), with swappable adhesives, as well as an app (Verily Patch app).

SUMMARY:
This is a single center, prospective, non-randomized prospective observational data collection study of the Verily Patch. The Verily Patch is an investigational wearable, continuous temperature sensor which will be evaluated against reference oral and axillary temperature measurements to support development activities for the Verily Patch.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Able to read and speak English
* Able to read and understand the Informed Consent Form
* Willing to wear Verily Patch in the axillary region
* Willing to comply with repeated self-measurement of oral and axillary temperatures and willing to record temperature readings
* Have a working smartphone device and willing to use it for study activities
* Willing to install study apps on their personal smartphone
* Willing to comply with all study-related procedures

Exclusion Criteria:

* Pregnant or breastfeeding during study participation
* Have known allergies to medical grade adhesives
* Have known cutaneous hypersensitivity
* Have infection in both axilla
* Have open injury or rash where the study device will be worn
* Have a cardiac pacemaker or other implanted electronic medical device(s)
* Have any additional condition or situation that, in the opinion of the investigator, makes the subject inappropriate for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 participants (50 febrile and 50 afebrile) will be enrolled at one investigational site. Febrile is defined as having sublingual temperatures of 37.50C or above. Participants that exhibit COVID-19 symptoms and/or COVID-19 diagnosis may be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Data collection to support development activities for Verily Patch | Up to 8 days
  Data collection to enable device development of the Verily Patch, which includes the development of an algorithm that estimates temperature

CONTACTS AND LOCATIONS:
Overall Officials: William Marks, MD, Study Director — Verily Life Sciences
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States